CLINICAL TRIAL: NCT03258164
Title: Fat Transplantation Enriched With Expanded Adipose-derived Autologous Mesenchymal Stromal Cells in Cosmetic Breast Augmentation and Cosmetic Facial Filling
Brief Title: Cosmetic Fat Transplantation Using Expanded ASC Enriched Fat Grafts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stemform (Industry)
Collaborators: Aleris-Hamlet Hospitaler København (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-16046960
Record Dates: First submitted 2017-08-07; First posted 2017-08-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Breast Hypoplasia and Facial Ageing

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC (Experimental)
  Interventions: Biological: ASC enriched lipofilling
- Control (Active Comparator)
  Interventions: Biological: Standard Lipofilling

INTERVENTIONS:
Biological: ASC enriched lipofilling — Fat grafts enriched with ex vivo expanded ASC
  Arms: ASC
Biological: Standard Lipofilling — Non-ASC enriched fat grafts
  Arms: Control

SUMMARY:
The purpose of the present study is to examine whether enrichment of a fat graft with autologous ex vivo expanded ASC injected into the breast tissue or face, both for cosmetic use, will significantly improve the results of conventional lipofilling and synthetic facial fillers, thereby being able to offer a safer, more natural and long-lasting alternative to current artificial solutions for cosmetic patients.

DETAILED DESCRIPTION:
The cosmetic breast augmentation design is a double-blind (surgeon and data assessor) randomized, prospective clinical study on healthy subjects.

The cosmetic facial filling design is a data assessor-blinded, randomized, prospective clinical study on healthy subjects.

ELIGIBILITY:
Criteria breast augmentation:

Inclusion criteria

1. Age 18 - 50 years
2. Healthy females
3. BMI 18 - 30 kg/m2
4. 1000 ml of fat (lipoaspirate) available for liposuction at the abdomen and/or thighs
5. Desire for breast augmentation
6. Speaks and reads Danish or English
7. Signed informed consent

Exclusion criteria

1. Smoking
2. Previous breast surgery
3. Previous cancer or predisposition to breast cancer
4. Pregnancy or planned pregnancy within one year after the procedure
5. Breastfeeding less than 6 months prior to inclusion
6. Weight gain or loss above 2 BMI point
7. Known chronic disease associated with metabolism malfunction or pour healing
8. Pacemaker or other implanted foreign objects
9. Allergy towards necessary anaesthesia
10. Intention of weight loss or weight gain within the trial period

Criteria fascial filling

Inclusion criteria

1. Age 25 - 65 years
2. Healthy females
3. BMI 18 - 30 kg/m2
4. 100 ml of fat (lipoaspirate) available for liposuction at the abdomen and/or thighs
5. Desire for facial wrinkle treatment and facial augmentation (rejuvenation)
6. Speaks and reads Danish or English
7. Signed informed consent

Exclusion criteria

1. Smoking
2. Previous facial surgery
3. Previous cancer
4. Pregnancy or planned pregnancy within one year after the procedure
5. Known chronic disease associated with metabolism malfunction or poor healing
6. Allergy towards necessary anaesthesia
7. Intention of weight loss or weight gain within the trial period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Change in volume over time after breast augmentation | Baseline, four and twelve months
  Measurement of the residual volume of fat transplants as based on MRI before operation (baseline), and four and twelve months after lipo-injection to the breast in order to determine the difference in volume between baseline and 4 months and 12 months post operative; and thereby the resorption rate over time.

SECONDARY OUTCOMES:
Change in cosmetic facial appearance over time after facial filling | Baseline, one, four and twelve months
  Assessment of cosmetic outcome based on clinical photos before (baseline), one, four and twelve months after the procedure when compared to baseline, evaluated by 5 independent plastic surgeons blinded to the intervention using a scale of 1-5 to determine the difference in appearance over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stig-Frederik T Kølle, MD, PhD, Principal Investigator — Stemform
Locations (1):
- Stemform, Copenhagen, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: No
Results will be published in international medical journals